CLINICAL TRIAL: NCT03719612
Title: A Phase III, Open-Label, Multicenter Trial to Evaluate Ejection Fraction, End-Diastolic and End-Systolic Volumes, by Unenhanced and DEFINITY®-Enhanced 2D-Echo and Magnetic Resonance Imaging
Brief Title: DEF-315 Better Accuracy in Ejection Fraction (EF) Assessment With DEFINITY
Acronym: BENEFIT2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lantheus Medical Imaging (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DEF-315
Record Dates: First submitted 2018-09-28; First posted 2018-10-25 (Actual); Results first posted 2021-01-07 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2019-11

CONDITIONS: Cardiac Disease
Keywords: Left Ventricular Ejection Fraction; DEFINITY®; Enhanced Echocardiogram; Cardiac Magnetic Resonance
MeSH Terms: conditions — Heart Diseases | interventions — perflutren

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DEFINITY® (Experimental): Each patient will undergo an unenhanced ultrasound examination and a DEFINITY® contrast-enhanced ultrasound
  Interventions: Drug: DEFINITY®

INTERVENTIONS:
Drug: DEFINITY® — All subjects will receive a single dose of DEFINITY®

SUMMARY:
This is a Phase 3, prospective, open-label, multicenter study to evaluate Left Ventricular Ejection Fraction (LVEF) measurement accuracy and reproducibility of DEFINITY® contrast-enhanced and unenhanced echocardiography as compared with non-contrast cardiac magnetic resonance imaging (CMR) used as the truth standard.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 18 years of age in sinus rhythm
2. Able to communicate effectively with trial personnel
3. LVEF measurements obtained via 2D Echo with or without contrast obtained within 6 months prior to enrollment (Day 0)
4. Has provided signed informed consent after receiving a verbal and written explanation of this clinical trial

Exclusion Criteria:

1. Female subjects who are pregnant or lactating. All women of child bearing potential [WOCBP] must have a negative urine pregnancy test at screening regardless of contraceptive use history.
2. Women of child-bearing potential are excluded unless they:

   1. are post-menopausal defined as amenorrhea ≥ 12 consecutive months, OR
   2. have undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy), OR
   3. have been using an adequate and medically approved method of contraception to avoid pregnancy for at least 1 month prior to DEFINITY® dose administration and be willing to continue using the same method for the duration of the study.
3. Current illness or pathology that would prevent undergoing investigational product administration due to a significant safety risk to the patient.
4. Uncontrolled arterial hypertension (defined as systolic blood pressure ≥ 200 mmHg or diastolic blood pressure ≥ 110 mmHg) or arterial hypotension (defined as systolic blood pressure ≤ 90 mmHg).
5. Unstable cardiovascular status defined as:

   1. myocardial infarction or unstable angina pectoris within 6 months prior to enrollment/DEFINITY® dose administration day
   2. transient ischemic attack or stroke within 3 months prior to DEFINITY® dose administration
   3. symptomatic valvular heart disease or moderate to severe stenotic valvular heart disease
   4. clinically significant congenital heart defects
   5. current uncontrolled cardiac arrhythmias causing symptoms or hemodynamic compromise
   6. acute pulmonary embolus or pulmonary infarction
   7. acute myocarditis or pericarditis
   8. acute aortic dissection
   9. atrial fibrillation
6. any major surgery within 4 weeks prior to screening
7. known contraindications to undergoing CMR (e.g. implanted pacemakers, cardioverter, defibrillators) or claustrophobia
8. participation in any investigational drug, device, or placebo study within 30 days prior to screening
9. known hypersensitivity to perflutren, or any of the excipients in DEFINITY®
10. prisoners or those who are subject to compulsory detention or involuntary incarceration for treatment of either a psychiatric or physical illness (e.g., infectious disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2018-12-28 (Actual); Primary Completion 2020-01-09 (Actual); Study Completion 2020-01-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Banner University of Arizona Medical Center, Tucson, Arizona
  - Cedars Sinai, Los Angeles, California
  - University of California-Irvine, Orange, California
  - UC San Diego, San Diego, California
  - Alfieri Cardiology, Wilmington, Delaware
  - Northwestern Medical Group, Chicago, Illinois
  - Indiana University, Bloomington, Indiana
  - Baptist Hospital, Paducah, Kentucky
  - Mercy Unit Hospital, Coon Rapids, Minnesota
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Oregon Health and Sciences University, Portland, Oregon
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Baylor Scott White Research Institute, Temple, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DEFINITY®
Started | 160
Completed | 148
Not Completed | 12

BASELINE CHARACTERISTICS:
Population: Baseline data are calculated based on Safety Population
Arm/Group | DEFINITY®
Number analyzed (Participants) | 160
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 106
  >=65 years | 54
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 105
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14
  Not Hispanic or Latino | 146
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 32
  White | 120
  More than one race | 2
  Unknown or Not Reported | 0
LVEF Group [Count of Participants; unit: Participants]
  LVEF <30% | 45
  LVEF 30-40% | 48
  LVEF 41-50% | 27
  LVEF >50% | 40

OUTCOME MEASURES:

1. Primary Outcome: Absolute Value of LVEF Percentage Differences From CMR by Blinded Reader
Description: Demonstrate improvement in accuracy in left ventricular ejection fraction (LVEF) assessment using DEFINITY® contrast-enhanced over unenhanced echocardiography by comparing LVEF percentage differences from CMR measured by 3 independent blinded image readers.
Time Frame: Up to 30 days between day of echocardiograms and CMR imaging
Population: Modified ITT Population
Measure: Mean (Standard Deviation); unit: Percent Ejection Fraction
Groups:
- Blinded Reader 1: Independent Blinded Reader 1 of 3
- Blinded Reader 2: Independent Blinded Reader 2 of 3
- Blinded Reader 3: Independent Blinded Reader 3 of 3
Arm/Group | Blinded Reader 1 | Blinded Reader 2 | Blinded Reader 3
Number analyzed (Participants) | 144 | 144 | 144
Percent Ejection Fraction
  Echo Enhanced | 5.70 (4.292) | 5.88 (4.330) | 5.03 (3.548)
  Echo Unenhanced | 6.08 (4.530) | 6.00 (4.813) | 5.36 (3.889)
Statistical Analysis 1: Comparison: Blinded Reader 1; Test type: Superiority — Difference between Echo Enhanced and Echo Unenhanced; p = 0.358, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = -0.38, Standard Deviation 4.947
Statistical Analysis 2: Comparison: Blinded Reader 2; Test type: Superiority — Difference between Echo Enhanced and Echo Unenhanced; p = 0.804, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = -0.12, Standard Deviation 5.699
Statistical Analysis 3: Comparison: Blinded Reader 3; Test type: Superiority — Difference between Echo Enhanced and Echo Unenhanced; p = 0.371, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = -0.33, Standard Deviation 4.412

2. Secondary Outcome: Secondary Objective 1: Absolute Value of LVEF Percentage Differences From CMR by Blinded Reader for Sub-optimal Echocardiograms
Description: Demonstrate improvement in accuracy in left ventricular ejection fraction (LVEF) assessment using DEFINITY® contrast-enhanced over unenhanced echocardiography in subjects with suboptimal echocardiograms by comparing LVEF percentage differences from CMR measured by 3 independent blinded readers.
Time Frame: Up to 30 days between day of echocardiogram and CMR imaging
Population: Modified ITT Population - Sub-optimal Echocardiograms
Measure: Mean (Standard Deviation); unit: Percent Ejection Fraction
Arm/Group | Blinded Reader 1 | Blinded Reader 2 | Blinded Reader 3
Number analyzed (Participants) | 48 | 48 | 48
Percent Ejection Fraction
  Echo Enhanced | 5.67 (3.717) | 6.16 (3.746) | 4.68 (3.456)
  Echo Unenhanced | 6.95 (5.219) | 6.81 (4.694) | 5.33 (3.764)
Statistical Analysis 1: Comparison: Blinded Reader 1; Test type: Superiority — Difference between Echo Enhanced and Echo Unenhanced; p = 0.030, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = -1.28, Standard Deviation 3.952
Statistical Analysis 2: Comparison: Blinded Reader 2; Test type: Superiority — Difference between Echo Enhanced and Echo Unenhanced; p = 0.312, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = -0.66, Standard Deviation 4.466
Statistical Analysis 3: Comparison: Blinded Reader 3; Test type: Superiority — Difference between Echo Enhanced and Echo Unenhanced; p = 0.347, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = -0.65, Standard Deviation 4.725

3. Secondary Outcome: Secondary Objective 2: Absolute Value LVEF Percentage Differences From CMR Between Blinded Readers
Description: Demonstrate a reduction in inter-reader variability for the assessment of left ventricular ejection fraction using DEFINITY® contrast-enhanced versus unenhanced echocardiography by comparing LVEF percentage differences from CMR between 3 independent blinded readers.
Time Frame: Up to 30 days between day of echocardiograms and CMR imaging
Population: Modified ITT Population
Measure: Mean (Standard Deviation); unit: Percent Ejection Fraction
Arm/Group | Blinded Reader 1 | Blinded Reader 2 | Blinded Reader 3
Number analyzed (Participants) | 144 | 144 | 144
Percent Ejection Fraction
  Echo Enhanced | 5.70 (4.292) | 5.88 (4.330) | 5.03 (3.548)
  Echo Unenhanced | 6.08 (4.530) | 6.00 (4.813) | 5.36 (3.889)
Statistical Analysis 1: Comparison: Blinded Reader 1 vs Blinded Reader 2; Inter-Reader Variability Echo Enhanced; Test type: Other; Intra-class Correlation Coefficient = 0.984, 95% CI 2-sided [0.977 to 0.988]
Statistical Analysis 2: Comparison: Blinded Reader 1 vs Blinded Reader 2; Inter-Reader Variability Echo Unenhanced; Test type: Other; Intra-class Correlation Coefficient = 0.953, 95% CI 2-sided [0.936 to 0.966]
Statistical Analysis 3: Comparison: Blinded Reader 1 vs Blinded Reader 3; Inter-Reader Variability Echo Enhanced; Test type: Other; Intra-class Correlation Coefficient = 0.970, 95% CI 2-sided [0.958 to 0.978]
Statistical Analysis 4: Comparison: Blinded Reader 1 vs Blinded Reader 3; Inter-Reader Variability Echo Unenhanced; Test type: Other; Intra-class Correlation Coefficient = 0.944, 95% CI 2-sided [0.923 to 0.959]
Statistical Analysis 5: Comparison: Blinded Reader 2 vs Blinded Reader 3; Inter-Reader Variability Echo Enhanced; Test type: Other; Intra-class Correlation Coefficient = 0.961, 95% CI 2-sided [0.947 to 0.972]
Statistical Analysis 6: Comparison: Blinded Reader 2 vs Blinded Reader 3; Inter-Reader Variability Echo Unenhanced; Test type: Other; Intra-class Correlation Coefficient = 0.942, 95% CI 2-sided [0.920 to 0.958]

4. Secondary Outcome: Secondary Objective 3: Absolute Value End-diastolic and Systolic Volume Differences From CMR Between Blinded Readers
Description: Demonstrate a reduction in inter-reader variability for the assessment of end-diastolic/systolic volumes using DEFINITY® contrast-enhanced versus unenhanced echocardiography by comparing end-diastolic and systolic volume differences from CMR between 3 independent blinded readers.
Time Frame: Up to 30 days between day of echocardiogram and CMR imaging
Population: Modified ITT Population
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Blinded Reader 1 | Blinded Reader 2 | Blinded Reader 3
Number analyzed (Participants) | 144 | 144 | 144
mL
  Echo Enhanced End Diastolic | 57.85 (44.204) | 51.13 (43.391) | 47.97 (40.589)
  Echo Unenhanced End Diastolic | 64.91 (44.084) | 62.01 (43.392) | 48.32 (39.895)
  Echo Enhanced End Systolic | 38.05 (32.921) | 32.41 (32.896) | 31.68 (30.603)
  Echo Unenhanced End Systolic | 42.87 (34.793) | 39.08 (34.139) | 32.45 (31.314)
Statistical Analysis 1: Comparison: Blinded Reader 1 vs Blinded Reader 2; Inter-Reader Variability End Diastolic Echo Enhanced; Test type: Other; Intra-class Correlation Coefficient = 0.984, 95% CI 2-sided [0.978 to 0.988]
Statistical Analysis 2: Comparison: Blinded Reader 1 vs Blinded Reader 2; Inter-Reader Variability End Diastolic Echo Unenhanced; Test type: Other; Intra-class Correlation Coefficient = 0.976, 95% CI 2-sided [0.967 to 0.983]
Statistical Analysis 3: Comparison: Blinded Reader 1 vs Blinded Reader 3; Inter-Reader Variability End Diastolic Echo Enhanced; Test type: Other; Intra-class Correlation Coefficient = 0.973, 95% CI 2-sided [0.963 to 0.981]
Statistical Analysis 4: Comparison: Blinded Reader 1 vs Blinded Reader 3; Inter-Reader Variability End Diastolic Echo Unenhanced; Test type: Other; Intra-class Correlation Coefficient = 0.935, 95% CI 2-sided [0.910 to 0.952]
Statistical Analysis 5: Comparison: Blinded Reader 2 vs Blinded Reader 3; Inter-Reader Variability End Diastolic Echo Enhanced; Test type: Other; Intra-class Correlation Coefficient = 0.973, 95% CI 2-sided [0.962 to 0.980]
Statistical Analysis 6: Comparison: Blinded Reader 2 vs Blinded Reader 3; Inter-Reader Variability End Diastolic Echo Unenhanced; Test type: Other; Intra-class Correlation Coefficient = 0.924, 95% CI 2-sided [0.896 to 0.945]
Statistical Analysis 7: Comparison: Blinded Reader 1 vs Blinded Reader 2; Inter-Reader Variability End Systolic Echo Enhanced; Test type: Other; Intra-class Correlation Coefficient = 0.989, 95% CI 2-sided [0.984 to 0.992]
Statistical Analysis 8: Comparison: Blinded Reader 1 vs Blinded Reader 2; Inter-Reader Variability End Systolic Echo Unenhanced; Test type: Other; Intra-class Correlation Coefficient = 0.983, 95% CI 2-sided [0.977 to 0.988]
Statistical Analysis 9: Comparison: Blinded Reader 1 vs Blinded Reader 3; Inter-Reader Variability End Systolic Echo Enhanced; Test type: Other; Intra-class Correlation Coefficient = 0.984, 95% CI 2-sided [0.978 to 0.989]
Statistical Analysis 10: Comparison: Blinded Reader 1 vs Blinded Reader 3; Inter-Reader Variability End Systolic Echo Unenhanced; Test type: Other; Intra-class Correlation Coefficient = 0.948, 95% CI 2-sided [0.928 to 0.962]
Statistical Analysis 11: Comparison: Blinded Reader 2 vs Blinded Reader 3; Inter-Reader Variability End Systolic Echo Enhanced; Test type: Other; Intra-class Correlation Coefficient = 0.978, 95% CI 2-sided [0.969 to 0.984]
Statistical Analysis 12: Comparison: Blinded Reader 2 vs Blinded Reader 3; Inter-Reader Variability End Systolic Echo Unenhanced; Test type: Other; Intra-class Correlation Coefficient = 0.942, 95% CI 2-sided [0.920 to 0.958]

5. Secondary Outcome: Secondary Objective 4: Absolute Value of LVEF Percentage Differences From CMR Between Readers for Sub-optimal Echocardiograms
Description: Demonstrate a reduction in inter-reader variability for the assessment of left ventricular ejection fraction using DEFINITY® contrast-enhanced versus unenhanced echocardiography by comparing LVEF percentage differences from CMR between 3 independent blinded readers in subjects with suboptimal echocardiograms.
Time Frame: Up to 30 days between day of echocardiograms and CMR imaging
Population: Modified ITT Population - Sub-optimal Echocardiograms
Measure: Mean (Standard Deviation); unit: Percent Ejection Fraction
Arm/Group | Blinded Reader 1 | Blinded Reader 2 | Blinded Reader 3
Number analyzed (Participants) | 48 | 48 | 48
Percent Ejection Fraction
  Echo Enhanced | 5.67 (3.717) | 6.16 (3.746) | 4.68 (3.456)
  Echo Unenhanced | 6.95 (5.219) | 6.81 (4.694) | 5.33 (3.764)
Statistical Analysis 1: Comparison: Blinded Reader 1 vs Blinded Reader 2; Inter-Reader Variability Echo Enhanced Sub-Optimal Echocardiograms; Test type: Other; Intra-class Correlation Coefficient = 0.975, 95% CI 2-sided [0.956 to 0.986]
Statistical Analysis 2: Comparison: Blinded Reader 1 vs Blinded Reader 2; Inter-Reader Variability Echo Unenhanced Sub-Optimal Echocardiograms; Test type: Other; Intra-class Correlation Coefficient = 0.936, 95% CI 2-sided [0.888 to 0.963]
Statistical Analysis 3: Comparison: Blinded Reader 1 vs Blinded Reader 3; Inter-Reader Variability Echo Enhanced Sub-Optimal Echocardiograms; Test type: Other; Intra-class Correlation Coefficient = 0.961, 95% CI 2-sided [0.931 to 0.978]
Statistical Analysis 4: Comparison: Blinded Reader 1 vs Blinded Reader 3; Inter-Reader Variability Echo Unenhanced Sub-Optimal Echocardiograms; Test type: Other; Intra-class Correlation Coefficient = 0.921, 95% CI 2-sided [0.864 to 0.955]
Statistical Analysis 5: Comparison: Blinded Reader 2 vs Blinded Reader 3; Inter-Reader Variability Echo Enhanced Sub-Optimal Echocardiograms; Test type: Other; Intra-class Correlation Coefficient = 0.947, 95% CI 2-sided [0.907 to 0.970]
Statistical Analysis 6: Comparison: Blinded Reader 2 vs Blinded Reader 3; Inter-Reader Variability Echo Unenhanced Sub-Optimal Echocardiograms; Test type: Other; Intra-class Correlation Coefficient = 0.903, 95% CI 2-sided [0.834 to 0.945]

6. Secondary Outcome: Secondary Objective 5: Absolute Value End-diastolic and Systolic Volume Differences From CMR Between Blinded Readers for Suboptimal Echocardiograms
Description: Demonstrate a reduction in inter-reader variability for the assessment of end-diastolic/systolic volumes using DEFINITY® contrast-enhanced versus unenhanced echocardiography by comparing end-diastolic and systolic volume differences from CMR between 3 independent blinded readers in subjects with suboptimal echocardiograms.
Time Frame: Up to 30 days between day of echocardiograms and CMR imaging
Population: Modified ITT Population - Sub-optimal Echocardiograms
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Blinded Reader 1 | Blinded Reader 2 | Blinded Reader 3
Number analyzed (Participants) | 48 | 48 | 48
mL
  Echo Enhanced End Diastolic | 71.67 (49.916) | 63.73 (49.571) | 61.86 (47.523)
  Echo Unenhanced End Diastolic | 74.89 (51.468) | 69.07 (46.316) | 64.38 (46.827)
  Echo Enhanced End Systolic | 45.59 (32.844) | 38.55 (33.493) | 39.52 (30.946)
  Echo Unenhanced End Systolic | 48.00 (37.639) | 41.88 (32.989) | 40.72 (32.333)
Statistical Analysis 1: Comparison: Blinded Reader 1 vs Blinded Reader 2; Inter-Reader Variability End Diastolic Echo Enhanced Sub-Optimal Echocardiograms; Test type: Other; Intra-class Correlation Coefficient = 0.984, 95% CI 2-sided [0.971 to 0.991]
Statistical Analysis 2: Comparison: Blinded Reader 1 vs Blinded Reader 2; Inter-Reader Variability End Diastolic Echo Unenhanced Sub-Optimal Echocardiograms; Test type: Other; Intra-class Correlation Coefficient = 0.975, 95% CI 2-sided [0.956 to 0.986]
Statistical Analysis 3: Comparison: Blinded Reader 1 vs Blinded Reader 3; Inter-Reader Variability End Diastolic Echo Enhanced Sub-Optimal Echocardiograms; Test type: Other; Intra-class Correlation Coefficient = 0.977, 95% CI 2-sided [0.959 to 0.987]
Statistical Analysis 4: Comparison: Blinded Reader 1 vs Blinded Reader 3; Inter-Reader Variability End Diastolic Echo Unenhanced Sub-Optimal Echocardiograms; Test type: Other; Intra-class Correlation Coefficient = 0.940, 95% CI 2-sided [0.896 to 0.966]
Statistical Analysis 5: Comparison: Blinded Reader 2 vs Blinded Reader 3; Inter-Reader Variability End Diastolic Echo Enhanced Sub-Optimal Echocardiograms; Test type: Other; Intra-class Correlation Coefficient = 0.977, 95% CI 2-sided [0.959 to 0.987]
Statistical Analysis 6: Comparison: Blinded Reader 2 vs Blinded Reader 3; Inter-Reader Variability End Diastolic Echo Unenhanced Sub-Optimal Echocardiograms; Test type: Other; Intra-class Correlation Coefficient = 0.923, 95% CI 2-sided [0.866 to 0.956]
Statistical Analysis 7: Comparison: Blinded Reader 1 vs Blinded Reader 2; Inter-Reader Variability End Systolic Echo Enhanced Sub-Optimal Echocardiograms; Test type: Other; Intra-class Correlation Coefficient = 0.990, 95% CI 2-sided [0.982 to 0.994]
Statistical Analysis 8: Comparison: Blinded Reader 1 vs Blinded Reader 2; Inter-Reader Variability End Systolic Echo Unenhanced Sub-Optimal Echocardiograms; Test type: Other; Intra-class Correlation Coefficient = 0.976, 95% CI 2-sided [0.957 to 0.986]
Statistical Analysis 9: Comparison: Blinded Reader 1 vs Blinded Reader 3; Inter-Reader Variability End Systolic Echo Enhanced Sub-Optimal Echocardiograms; Test type: Other; Intra-class Correlation Coefficient = 0.985, 95% CI 2-sided [0.973 to 0.991]
Statistical Analysis 10: Comparison: Blinded Reader 1 vs Blinded Reader 3; Inter-Reader Variability End Systolic Echo Unenhanced Sub-Optimal Echocardiograms; Test type: Other; Intra-class Correlation Coefficient = 0.929, 95% CI 2-sided [0.876 to 0.959]
Statistical Analysis 11: Comparison: Blinded Reader 2 vs Blinded Reader 3; Inter-Reader Variability End Systolic Echo Enhanced Sub-Optimal Echocardiograms; Test type: Other; Intra-class Correlation Coefficient = 0.981, 95% CI 2-sided [0.966 to 0.989]
Statistical Analysis 12: Comparison: Blinded Reader 2 vs Blinded Reader 3; Inter-Reader Variability End Systolic Echo Unenhanced Sub-Optimal Echocardiograms; Test type: Other; Intra-class Correlation Coefficient = 0.916, 95% CI 2-sided [0.855 to 0.952]

ADVERSE EVENTS:
Time Frame: Up to 12 days: Enrolled subjects were followed for adverse events and serious adverse events from the time the Informed Consent was signed at screening (Day -7 to Day 0) through 72+/-24 hours after completion of Definity administration (Day 0).
Arm/Group | DEFINITY®
All-Cause Mortality (participants affected / at risk) | 0/160
Serious Adverse Events (participants affected / at risk) | 1/160
Other Adverse Events (participants affected / at risk) | 0/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DEFINITY® (N=160)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-15): https://cdn.clinicaltrials.gov/large-docs/12/NCT03719612/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-31): https://cdn.clinicaltrials.gov/large-docs/12/NCT03719612/SAP_001.pdf